CLINICAL TRIAL: NCT06480552
Title: A Phase 1a/1b Open-Label, Multicenter, Dose Escalation, and Dose Expansion Trial to Evaluate the Safety and Activity of TEV-56278, as a Monotherapy and in Combination With Pembrolizumab in Participants With Selected Locally Advanced or Metastatic Solid Tumors
Brief Title: An Open-label Dose Escalation/Expansion Trial to Evaluate the Safety and Anti-tumor Activity of TEV-56278 Alone or in Combination With Pembrolizumab in Participants With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TV56278-ONC-10203
Record Dates: First submitted 2024-06-10; First posted 2024-06-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TEV-56278 Monotherapy; Dose Escalation (Experimental)
  Interventions: Drug: TEV-56278
- TEV-56278 Monotherapy; Dose Expansion (Experimental)
  Interventions: Drug: TEV-56278
- TEV-56278 in Combination with Pembrolizumab; Dose Escalation (Experimental)
  Interventions: Drug: TEV-56278; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TEV-56278 — Administered intravenously
Drug: Pembrolizumab — Administered intravenously
  Other Names: KEYTRUDA®
  Arms: TEV-56278 in Combination with Pembrolizumab; Dose Escalation

SUMMARY:
The primary objectives of this trial are to:

* Characterize the safety and tolerability of TEV-56278
* Determine the Recommended Phase 2 Dose (RP2D)
* Evaluate antitumor activity of TEV-56278
* Determine the safety and tolerability of TEV-56278 in combination with pembrolizumab
* Determine a RP2D of TEV-56278 in combination with pembrolizumab

The secondary objectives of this trial are to:

* Characterize the serum pharmacokinetics of TEV-56278
* Evaluate the antitumor activity of TEV-56278
* Determine the safety and tolerability of TEV-56278
* Evaluate other measures of antitumor activity of TEV-56278
* Evaluate anti-tumor activity

Participants will be treated up to 12 months with a follow-up period of up to 12 months after last infusion. The total duration of the trial will be up to 25 months for individual participants.

ELIGIBILITY:
Inclusion Criteria:

* Have an established histological diagnosis of selected solid tumor and must have received and progressed on established standard therapies or have been intolerant to such therapy or have been considered by the Investigator as ineligible for approved standard therapy
* Have a life expectancy≥12 weeks at the time of the screening
* Women of childbearing potential must agree to use highly effective methods of contraception for the course of the trial through 120 days after the last dose of trial medication
* Males who are sexually active with women of childbearing potential must agree to use condoms and refrain from donating sperm for the course of the trial through 120 days after the last dose of trial medication

NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Has a history of systemic treatment therapy for cancer (including chemotherapy, immunotherapy, radiotherapy, or other investigational drug) or surgery within 4 weeks prior to baseline
* Is currently receiving or has received hematopoietic colony-stimulating growth factors within 2 weeks before screening or transfusion support 4 weeks prior to screening
* Has a diagnosis of immunodeficiency
* Has active known autoimmune disease.
* Has a history of or known active brain metastases and/or carcinomatous meningitis and/or leptomeningeal metastasis
* Has active or uncontrolled serious infections requiring systemic therapy within 14 days prior to baseline
* Has a history of clinically significant cardiovascular or cerebrovascular disease in previous 6 months prior to screening
* Has evidence of clinically significant interstitial lung disease or active, noninfectious pneumonitis
* Has a seizure disorder requiring therapy (such as steroids or antiepileptics)

NOTE- Additional criteria apply, please contact the investigator for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2029-05-26 (Estimated); Study Completion 2031-02-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs with CTCAE Grade≥3 in the escalation phase | Up to 15 months after 1st infusion in the escalation phase
  CTCAE: Common Terminology Criteria for Adverse Events
Incidence of SAEs in the escalation phase | Up to 15 months after 1st infusion in the escalation phase
Incidence of AEs meeting protocol-defined DLT criteria in the escalation phase | Up to 28 days after 1st infusion in the escalation phase
  DLT: dose-limiting toxicity
Incidence of dose modifications due to AEs in the escalation phase | Up to 12 months after 1st infusion in the escalation phase
Incidence of AEs leading to discontinuation in the escalation phase | Up to 12 months after 1st infusion in the escalation phase
Recommended Phase 2 dose as monotherapy | Up to 24 months after 1st infusion
Objective Response Rate (ORR) based on RECIST criteria in the expansion phase | Up to 24 months after the 1st dose in the expansion phase
  RECIST: Response Evaluation Criteria in Solid Tumors.
Duration of Response (DOR) in the expansion phase | Up to 24 months after the 1st dose in the expansion phase
Recommended Phase 2 dose in combination with Pembrolizumab | Up to 24 months after 1st dose
Incidence of AEs with CTCAE Grade≥3 in the combination phase | Up to 15 months after 1st infusion in the combination phase
Incidence of SAEs in the combination phase | Up to 15 months after 1st infusion in the combination phase
Incidence of AEs meeting protocol-defined DLT criteria in the combination phase | Up to 28 days after 1st infusion in the combination phase
Incidence of dose modifications due to AEs in the combination phase | Up to 12 months after 1st infusion in the combination phase
Incidence of AEs leading to discontinuation in the combination phase | Up to 12 months after 1st infusion in the combination phase

SECONDARY OUTCOMES:
AUC0-last | Predose up to Day 8
  Area under the serum concentration-time curve from time 0 to last measurable drug concentration
Cmax | Predose up to Day 8
  Maximum observed concentration
tmax | Predose up to Day 8
  Time to maximum observed drug concentration
Objective Response Rate (ORR) based on RECIST criteria in the escalation phase | Up to 24 months after 1st infusion in the escalation phase
Incidence of AEs with CTCAE Grade≥3 in the expansion phase | Up to 24 months after 1st infusion in the expansion phase
Incidence of SAEs in the expansion phase | Up to 15 months after 1st infusion in the expansion phase
Incidence of dose modifications due to AEs in the expansion phase | Up to 12 months after 1st infusion in the expansion phase
Incidence of AEs leading to discontinuation in the expansion phase | Up to 12 months after 1st infusion in the expansion phase
Disease Control Rate (DCR) according to RECIST (v1.1) criteria | Up to 24 months after 1st infusion
Time to Respond (TTR) according to RECIST (v1.1) criteria | Up to 24 months after 1st infusion
Objective Response Rate (ORR) based on RECIST criteria in the combination phase | Up to 24 months after 1st infusion in the combination phase

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (11):
- United States (10):
  - Teva Investigational Site 12017, Los Angeles, California
  - Teva Investigational Site 12021, Lake Mary, Florida
  - Teva Investigational Site 12016, Chicago, Illinois
  - Teva Investigational Site 12015, Detroit, Michigan
  - Teva Investigational Site 12014, Huntersville, North Carolina
  - Teva Investigational Site 12023, Cincinnati, Ohio
  - Teva Investigational Site 12058, Pittsburgh, Pennsylvania
  - Teva Investigational Site 12019, Nashville, Tennessee
  - Teva Investigational Site 12018, Fairfax, Virginia
  - Teva Investigational Site 12025, Milwaukee, Wisconsin
- Teva Investigational Site 11282, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.